CLINICAL TRIAL: NCT01720667
Title: Efficacy of Intravenous Levetiracetam in Neonatal Seizures: A Phase 2 Randomized Blinded Controlled Study of the Efficacy of Intravenous Levetiracetam (LEV) as First Line Treatment for Neonatal Seizures
Brief Title: Efficacy of Intravenous Levetiracetam in Neonatal Seizures
Acronym: NEOLEV2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Richard H. Haas (Other)
Collaborators: University of California, San Diego (Other); Rady Children's Hospital, San Diego (Other); Auckland City Hospital (Other Government); Sharp Mary Birch Hospital for Women & Newborns (Other); UCSF Benioff Children's Hospital Oakland (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Richard H. Haas, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NoGA - R01 FD004147-01A1 Haas; 1R01FD004147-01A1 (FDA)
Record Dates: First submitted 2012-10-22; First posted 2012-11-02 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Neonatal Seizures
Keywords: Seizures; Neonates; Anticonvulsants; Treatment; Levetiracetam; Phenobarbital
MeSH Terms: conditions — Seizures | interventions — Levetiracetam; Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous levetiracetam (Experimental): Intravenous levetiracetam 40 to 60 mg/kg loading dose. 10 mg/kg 8 hourly maintenance
  Interventions: Drug: Intravenous levetiracetam
- Intravenous phenobarbital (Active Comparator): Intravenous phenobarbital 20 to 40 mg/kg load. 1.5 mg/kg 8 hourly maintenance
  Interventions: Drug: Intravenous phenobarbital

INTERVENTIONS:
Drug: Intravenous levetiracetam — Intravenous load of levetiracetam (40 to 60 mg/kg) following identification of EEG confirmed neonatal seizure.
  Other Names: Keppra
  Arms: Intravenous levetiracetam
Drug: Intravenous phenobarbital — Intravenous load of phenobarbital (20 to 40 mg/kg) following EEG confirmation of seizure activity load.
  Other Names: phenobarbitone
  Arms: Intravenous phenobarbital

SUMMARY:
A new anticonvulsant, levetiracetam will be studied to treat seizures in newborn infants. Current treatments for the brain damaging complication of neonatal seizures are unsatisfactory.

Monitoring for seizure detection will be tested at five (5) US sites and one (1) international site using the internet.

DETAILED DESCRIPTION:
This project aims to improve the treatment of neonatal seizures. Current treatments are poorly effective and have significant side effects.

Levetiracetam (LEV) has great potential as a treatment for neonatal seizures but is not approved for use in children less than 2 years of age.

This study aims to obtain essential data regarding the efficacy and safety of LEV in this vulnerable and under researched population and simultaneously to develop EEG monitoring systems that facilitate seizure detection and research.

Specific aims are:

1. To determine the efficacy of intravenous LEV in terminating neonatal seizures when given as first line therapy.
2. To obtain dose escalation data by studying the additional efficacy of a further dose in non responders.
3. To obtain additional pharmacokinetic data to confirm findings from our previous pharmacokinetic study.
4. To obtain further safety data of LEV in neonates.
5. To prove the feasibility of centralized remote monitoring of continuous EEG monitoring in the Neonatal Intensive Care Unit (NICU) via the internet and test a promising automated neonatal seizure detection algorithm.

The study design is a phase 2b randomized blinded controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns admitted to any of the study sites with electrographic seizures seizures.
2. Term infants gestational age >36 weeks less than 2 weeks of age.
3. Greater than 2200 grams.
4. Infants for whom parental consent to participate in the study is obtained.

Exclusion Criteria:

1. Infants who are already receiving anticonvulsants
2. If serum creatinine is greater than 1.6mM
3. If seizures are due to correctable metabolic abnormalities (i.e. hypoglycaemia, hypocalcemia, hyponatremia)
4. Subjects in whom death seems imminent, as assessed by the neonatologist.

Ages: 15 Minutes to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Haas, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Medical Center / Neonatal Intensive Care Unit (NICU), San Diego, California, United States

REFERENCES:
- [Background] Sharpe CM, Capparelli EV, Mower A, Farrell MJ, Soldin SJ, Haas RH. A seven-day study of the pharmacokinetics of intravenous levetiracetam in neonates: marked changes in pharmacokinetics occur during the first week of life. Pediatr Res. 2012 Jul;72(1):43-9. doi: 10.1038/pr.2012.51. Epub 2012 Apr 11. PMID 22495532
- [Result] Sharpe C, Davis SL, Reiner GE, Lee LI, Gold JJ, Nespeca M, Wang SG, Joe P, Kuperman R, Gardner M, Honold J, Lane B, Knodel E, Rowe D, Battin MR, Bridge R, Goodmar J, Castro B, Rasmussen M, Arnell K, Harbert M, Haas R. Assessing the Feasibility of Providing a Real-Time Response to Seizures Detected With Continuous Long-Term Neonatal Electroencephalography Monitoring. J Clin Neurophysiol. 2019 Jan;36(1):9-13. doi: 10.1097/WNP.0000000000000525. PMID 30289769
- [Derived] Sharpe C, Yang DZ, Haas RH, Reiner GE, Lee L, Capparelli EV; NEOLEV2 Investigators. Pharmacokinetic and pharmacodynamic data from the NEOLEV1 and NEOLEV2 studies. Arch Dis Child. 2024 Sep 25;109(10):854-860. doi: 10.1136/archdischild-2022-324952. PMID 38902005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 280 were enrolled to EEG monitoring and of these 106 were randomized to treatment as neonatal seizures were thought to have occurred. 174 excluded as they did not have electrographic seizures; from 6 participants only verbal not written consent obtained.
Groups:
- Intravenous Levetiracetam: Intravenous levetiracetam 40 - 60 mg/kg loading dose. If electrographic seizures persisted or recurred 15 minutes following completion of the infusion, subjects received a further 20 mg/kg LEV infusion over 15 minutes. If electrographic seizures persisted or recurred 15 minutes following completion of the second infusion, the subject was then treated with PHB 20 mg/kg. Another dose of 20 mg/kg PHB given if seizures persist. Unresponsive subjects exit the study. All subjects received maintenance LEV 10 mg/kg/dose given IV q8 hours continued for five days.
- Intravenous Phenobarbital: Intravenous phenobarbital 20 mg/kg loading dose. If electrographic seizures persisted or recurred 15 minutes following completion of the infusion, subjects received a further 20 mg/kg PHB infusion over 15 minutes. If electrographic seizures persisted or recurred 15 minutes following completion of the second infusion, the subject was then treated with LEV 40 mg/kg first. Another dose of 20 mg/kg PHB given if seizures persist. Unresponsive subjects exit the study. All subjects received maintenance 1.5 mg/kg PHB mg/kg/dose given IV q8 hours continued for five days.
Period: Overall Study
Arm/Group | Intravenous Levetiracetam | Intravenous Phenobarbital
Started | 64 | 42
Recieved Second Infusion of Same Drug | 50 | 20
Recieved Alternate Intervention | 45 | 10
Received 2nd Infusion of Alternate Drug | 27 | 6
Modified ITT | 53 | 30
Completed | 60 | 41
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Levetiracetam | Intravenous Phenobarbital | Total
Number analyzed (Participants) | 64 | 42 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 42 | 106
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 18 | 51
  Male | 31 | 24 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 10 | 28
  Not Hispanic or Latino | 39 | 25 | 64
  Unknown or Not Reported | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 7 | 2 | 9
  Black or African American | 4 | 1 | 5
  White | 34 | 25 | 59
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 45 | 30 | 53
  New Zealand | 19 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Neonates With Seizure Cessation When Given Levetiracetam (40-60 mg/kg) as First Line Therapy Compared to Phenobarbital (20-40mg/kg)
Description: A head to head comparison of the efficacy of intravenous levetiracetam versus phenobarbital in the treatment of EEG proven neonatal seizures.
  Seizure cessation from 15 minutes after completion of infusion for 24 hours as assessed by continuous EEG reviewed by neurophysiologists.
Time Frame: 24 hours
Population: Treated participants with available primary outcome measure- EEG to 24 hours confirming seizure cessation.
Measure: Count of Participants; unit: Participants
Groups:
- Intravenous Levetiracetam: Intravenous levetiracetam 40 - 60 mg/kg loading dose & 10 mg/kg 8 hourly maintenance
- Intravenous Phenobarbital: Intravenous phenobarbital 20 - 40 mg/kg loading dose & 1.5 mg/kg 8 hourly maintenance.
Arm/Group | Intravenous Levetiracetam | Intravenous Phenobarbital
Number analyzed (Participants) | 53 | 30
Participants | 15 | 24
Statistical Analysis 1: Comparison: Intravenous Levetiracetam vs Intravenous Phenobarbital; Comparison of 24 hour seizure termination rates using a Fisher's exact test; Test type: Superiority; p < 0.001, Fisher Exact

2. Secondary Outcome: Neonates With Seizure Cessation When Given Levetiracetam as First Line Therapy Compared to Phenobarbital at 48 Hours After Treatment
Description: A head to head comparison of the efficacy of intravenous levetiracetam versus phenobarbital in the treatment of EEG proven neonatal seizures.
Time Frame: 48 hours
Population: Participants with evaluable data with 48 hours of seizure monitoring
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Levetiracetam | Intravenous Phenobarbital
Number analyzed (Participants) | 47 | 28
Participants | 8 | 18
Statistical Analysis 1: Comparison: Intravenous Levetiracetam vs Intravenous Phenobarbital; Comparison of seizure cessation at 48 hours using Fisher's exact test; Test type: Superiority; p < 0.001, Fisher Exact

3. Secondary Outcome: Number of Neonates With Seizure Termination at 1 Hour After Treatment
Description: as for outcome 2
Time Frame: 1 hour
Population: Includes 1 participant in each arm who did not have data available for the primary end point at 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Levetiracetam | Intravenous Phenobarbital
Number analyzed (Participants) | 53 | 30
Participants | 26 | 28

4. Secondary Outcome: LEV Dose Escalation Component
Description: Number of babies with seizure control at levetiracetam (60 mg/Kg load) who had not responded to 40 mg/kg load and number of babies with seizure control at 40 mg/kg who had not responded to 20 mg/kg.
Time Frame: 24 hours
Population: Babies who received any treatment of either phenobarbital or levetiracetam within the modified intent to treat
Measure: Count of Participants; unit: Participants
Groups:
- Intravenous Levetiracetam: Intravenous levetiracetam 40 mg/kg loading dose & 10 mg/kg 8 hourly maintenance
- Intravenous Phenobarbital: Intravenous phenobarbital 20 mg/kg loading dose & 1.5 mg/kg 8 hourly maintenance.
Arm/Group | Intravenous Levetiracetam | Intravenous Phenobarbital
Number analyzed (Participants) | 53 | 30
Participants | 4 | 3

5. Secondary Outcome: Neonates With Seizure Cessation When Given Levetiracetam as First Line Therapy Compared to Phenobarbital Within the Hypoxic Ischemic Encephalopathy (HIE) Population and Treated With Hypothermia
Time Frame: 24 hours
Population: HIE participants with hypothermia treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Levetiracetam | Intravenous Phenobarbital
Number analyzed (Participants) | 17 | 10
Participants | 6 | 9

6. Other Pre Specified Outcome: Pharmacokinetic Data
Description: To obtain additional pharmacokinetic data "Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax)" of intravenous levetiracetam to confirm findings from our previous pharmacokinetic study.
Time Frame: 48 hours
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Feasibility of Continuous Internet EEG Monitoring
Description: Feasibility of centralized remote access to continuous video EEG monitoring in the NICU via the internet
Time Frame: Subject study duration
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Evaluation of the Accuracy of Neonatal Seizure Detection Algorithm
Description: A novel neonatal seizure detection algorithm will be compared to the gold standard of two encephalographers reading 48 hours of neonatal video EEG in the measurement of seizure burden.
Time Frame: 48 Hours
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Gather Safety Information on IV Levetiracetam
Description: Safety information to be collected includes daily recording of any adverse events during the 5 day treatment protocol.
  Complete Blood Count and Comprehensive Chemistry panels after 48 hours of treatment collected.
Time Frame: 5 days
Reporting Status: Not Posted, anticipated posting 2019-09

10. Post Hoc Outcome: Imputation Sensitivity Analysis
Description: Analysis of missing data impact on the outcome measures
Time Frame: 48 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 days after treatment
Description: Data not collected separately for each intervention
Arm/Group | Intravenous Phenobarbital | Intravenous Levetiracetam
All-Cause Mortality (participants affected / at risk) | 1/42 | 2/64
Serious Adverse Events (participants affected / at risk) | 5/42 | 1/64
Other Adverse Events (participants affected / at risk) | 13/42 | 12/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Phenobarbital (N=42) | Intravenous Levetiracetam (N=64)
Hypotension (Vascular disorders) | 4 | 1 — Grade 4 hypotension thought probably or possibly due to study medications
Respiratory Abnormality (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Grade 4 respiratory distress thought probably or possibly due to study medication
Heart Rate Abnormality (Cardiac disorders) | 0 | 0
Sedation (Nervous system disorders) | 0 | 0
Poor Feeding (Gastrointestinal disorders) | 0 | 0
Infection (Infections and infestations) | 0 | 0
New Medications (General disorders) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Phenobarbital (N=42) | Intravenous Levetiracetam (N=64)
Hypotension (Vascular disorders) | 7 | 3 — Specific finding of hypotension on a day on which an adverse event was indicated.
Heart Rate Abnormailty (Cardiac disorders) | 1 | 3 — Specific finding of heart rate abnormality on a day on which an adverse event was reported
Respiratory Abnormality (Respiratory, thoracic and mediastinal disorders) | 12 | 8 — Specific finding of respiratory abnormality documented on a day on which an adverse event was documented
Sedation (Nervous system disorders) | 8 | 7 — Specific finding of sedation on a day on which an adverse event was documented
Poor Feeding (Gastrointestinal disorders) | 7 | 6 — Specific finding of poor feeding on a day on which adverse event was documented
Infection (Infections and infestations) | 3 | 2 — Specific finding of infection on a day on which adverse event was documented
New Medical Problem (General disorders) | 6 | 5 — New Medical Problem reported on a day where an adverse event is documented
New Medications (General disorders) | 7 | 3
Vasopressor Requirement (Cardiac disorders) | 13 (13) | 10 (10) — Hypotension requiring vasopressor support on at least one day

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT01720667/SAP_000.pdf
  • Study Protocol (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT01720667/Prot_001.pdf